CLINICAL TRIAL: NCT02779725
Title: SymptomCare@Home (SCH): Deconstructing an Effective, Technology-assisted, Symptom Management Intervention
Brief Title: SymptomCare@Home: Deconstructing an Effective Symptom Management Intervention
Acronym: SCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Huntsman Cancer Institute (Other); Emory University (Other)
Responsible Party: Principal Investigator, Kathleen Mooney, Distinguished Professor/Principal Investigator, University of Utah
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00087666; R01CA206522 (NIH)
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Cancer
Keywords: Symptom Management
MeSH Terms: conditions — Neoplasms | interventions — Nurse Practitioners; Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 SCC/SSR (Active Comparator): This arm includes self-care coaching (SCC) message during daily self-reported symptom severity report (SSR) calls to the automated system.
  Interventions: Behavioral: SCC; Behavioral: Symptom Severity
- Group 2 NP/SSR (Active Comparator): Alert reports are generated during the patient's daily symptom severity monitoring call if alert thresholds are reached. These alerts are monitored and follow-up care is given by a nurse practitioner.
  Interventions: Behavioral: Nurse Practitioner; Behavioral: Symptom Severity
- Group 3 NP/DSS/SSR (Active Comparator): Alert reports are generated during the patient's daily symptom severity monitoring call if alert thresholds are reached. Nurse practitioner follow-up calls utilize the evidenced based SCH decision support system (DSS) when symptoms exceed alert thresholds
  Interventions: Behavioral: Nurse Practitioner; Behavioral: DSS; Behavioral: Symptom Severity
- Group 4 Full Intervention SSR/SCC/NP/DSS (Active Comparator): Complete intervention with all components used in prior efficacy study (Symptom Severity Report (SSR)+Self Care Coaching (SCC) +Nurse Practitioner (NP) +Decision Support System (DSS))
  Interventions: Behavioral: SCC; Behavioral: Nurse Practitioner; Behavioral: DSS; Behavioral: Symptom Severity
- Group 5 SSR/SCC/AT (Active Comparator): Symptom severity reporting (SSR), automated self-care coaching (SCC) based on daily symptom reporting plus activity tracker (AT)
  Interventions: Behavioral: SCC; Behavioral: AT; Behavioral: Symptom Severity

INTERVENTIONS:
Behavioral: SCC — Automated self-management coaching paired to symptom reports during daily symptom monitoring call
  Other Names: Self-Management Coaching
  Arms: Group 1 SCC/SSR; Group 4 Full Intervention SSR/SCC/NP/DSS; Group 5 SSR/SCC/AT
Behavioral: Nurse Practitioner — Alerts generate if a patient reports symptoms above pre-set thresholds during daily symptom reporting calls . These alerts are monitored and follow up is given by a Nurse Practitioner.
  Other Names: Nurse Practitioner Follow Up
  Arms: Group 2 NP/SSR; Group 3 NP/DSS/SSR; Group 4 Full Intervention SSR/SCC/NP/DSS
Behavioral: DSS — A Clinical Decision Support System (DSS), based on evidenced based guidelines, will be used to assist the nurse practitioner in follow up to symptom alerts.
  Other Names: Clinical Decision Support System
  Arms: Group 3 NP/DSS/SSR; Group 4 Full Intervention SSR/SCC/NP/DSS
Behavioral: AT — An activity tracker will be provided to evaluate its use, acceptability and impact on fatigue severity. The purpose of providing the activity tracker is to extend the self-management coaching intervention given when participants report fatigue and receive coaching about exercise as part of the intervention.
  Other Names: Activity Tracker
  Arms: Group 5 SSR/SCC/AT
Behavioral: Symptom Severity — Automated patient-reporting of 11 common cancer treatment symptoms
  Other Names: Patient Reported Symptom Severity

SUMMARY:
This project will determine the most important and cost effective components of SymptomCare@Home, a new approach to cancer chemotherapy symptom care that has been shown to reduce problematic symptoms through automated daily monitoring, self-management coaching, and oncology team follow-up care using decisional support for patients at home when their symptoms are most likely at their worse. Once the key parts of the intervention and its cost effectiveness are known, it can be moved into everyday cancer care.

DETAILED DESCRIPTION:
Cancer patients receiving chemotherapy experience multiple poorly controlled symptoms at home in the interim weeks between clinic visits and the next infusion. Their care during this interim time period is suboptimal. Technology can be utilized to bridge the gap between patient symptom needs at home and oncology team response. Automated patient-reported symptom home monitoring and management systems offer a new approach to symptom care. Our research team has developed and tested SymptomCare@Home (SCH). This multi-component automated system monitors daily patient-reported symptoms at home, provides tailored automated self-management coaching based on the specific symptoms reported and transmits unrelieved symptom alert reports to an oncology provider who, using the SCH decision support system provides follow-up telephone-delivered symptom care. We have demonstrated that SCH dramatically reduces physical and psychological symptom severity. However there remain several gaps in translating a successful, multi-component symptom intervention into clinical practice. These include understanding 1) the contribution and value of each part of the intervention so that the active components are selected for clinical implementation and 2) the costs associated with the intervention and its components. Therefore the aims of this project are to deconstruct the SCH symptom monitoring and management system to determine the relative contribution and costs of its components to achieving symptom reduction, maintain general health functioning and reduce healthcare utilization. We will also examine who benefits most and least from the individual components and from the overall system. A 5 group randomized control trial design will be utilized with 750 participants (150/group) beginning a new course of chemotherapy who will call the SCH system daily and report the presence and severity of 11 symptoms throughout a course of chemotherapy or up to 6 months. This study is both significant and innovative because it shifts the current clinical practice paradigm for providing symptom care episodically during clinic visits to an innovative approach that is patient-centric, providing symptom care when and where the patient needs it. The study will address questions not generally asked in multi-component interventions, determining the active ingredients and their costs. Determining the value of new approaches to care such as automated telehealth interventions is essential to the decision process of healthcare systems and payers who decide what to adopt and reimburse. It is also vitally important to patients so that new symptom care innovations are adopted that better meet their needs and dramatically reduce their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of cancer
* Life expectance of at least three months
* Beginning a new course of chemotherapy that is planned for a minimum of three cycles
* English speaking
* Daily access to a telephone
* Cognitively capable to use the phone unassisted as verified by study staff at recruitment
* Receiving care under the direction of one of the designated provider teams at Huntsman Cancer Institute (SLC, UT) or Grady Cancer Institute (Atlanta, GA).

Exclusion Criteria:

* Receiving concurrent radiation therapy
* Exclusively receiving biotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 884 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Patient reported symptom levels | up to 6 months
  During daily automated calls, patients provided information about common chemotherapy symptoms on a 0-10 scale.

SECONDARY OUTCOMES:
Overall Health functioning: physical, mental, and social | up to 6 months
  This will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 + 2 items from the PROMIS 10 (92-95)
Work Interference | up to 6 months
  For patients who indicated they worked during their treatment, the system asked daily if they missed work if it was a regular workday.
Work Limitations Questionnaire | up to 6 months
  The 25 item patient-reported Work Limitations Questionnaire will be used to measure work performance.
Health Care Utilization & Medical Encounters Interview | up to 6 months
  Each week patients reported during their daily phone calls whether or not they had been in contact with a health care provider, were seen in an emergency department or urgent care facility, or had an unscheduled hospitalization. If they reported they did have a medical encounter, the research staff would call and conduct a short telephone interview to collect data about the nature of the medical encounter including whether the medical encounter was related to the symptoms being monitored.
Baseline Physical Activity | Baseline
  We will measure baseline physical activity using the 3 item Godin's Leisure-Time Exercise Questionnaire

OTHER OUTCOMES:
Patient End of Study Telephone Interview | up to 6 months
  An End of Study Telephone Interview will be conducted at the end of a patient's participation in the project to obtain data on patient satisfaction with the symptom monitoring system and to obtain suggestions for improvement of the system.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Mooney, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
We will present our findings at conferences and publish the findings. We welcome analysis and use by other investigators once our primary aims have been analyzed and disseminated. The PI will share de-identified data to other investigators for study, including demographics, diagnosis, chemotherapy treatment, symptom patterns, work attendance, overall health function and health care utilization. Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and can be used for secondary study purposes. The PI agrees to make available data within one year of the completion of the funded project period and manuscripts pertaining to the aims. De-identified data will be available directly from the PI. The PI agrees to share data in a manner that is fully consistent with NIH data sharing policies and applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available once the primary aims of the R01 study have been published.
Access Criteria: Data will be available to address research questions/hypothesis of the request. Once the Principal Investigator reviews the research question proposed, the data elements that can address the question will be shared.

REFERENCES:
- [Derived] Mooney K, Gullatte M, Iacob E, Alekhina N, Nicholson B, Sloss EA, Lloyd J, Moraitis AM, Donaldson G. Essential Components of an Electronic Patient-Reported Symptom Monitoring and Management System: A Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2433153. doi: 10.1001/jamanetworkopen.2024.33153. PMID 39269704

DOCUMENTS (1):
  • Informed Consent Form (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT02779725/ICF_000.pdf